CLINICAL TRIAL: NCT01480271
Title: A Randomized, Double-blind, Placebo-controlled First Time Into Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intranasal Dosing With GSK2245035, a TLR7 Agonist, in Healthy Volunteers and Allergic Rhinitics
Brief Title: An Investigation of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2245035 in Healthy Volunteers and Allergic Rhinitics.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114450
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Allergic Rhinitis; Healthy Volunteers; Single Dose Escalation; TLR7 agonist; First Time in Human Study
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- Part 1 Cohort 1 GSK2445053 (Experimental): 2ng GSK2245053
  Interventions: Drug: 2 ng GSK2445053
- Part 1 Cohort 1 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 2 GSK2445053 (Experimental): 20ng GSK2445053
  Interventions: Drug: 20ng GSK2445053
- Part 1 Cohort 2 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 3 GSK2245053 (Experimental): 100ng GSK2445053
  Interventions: Drug: 100ng GSK2445053
- Part 1 Cohort 3 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 4 GSK2445053 (Experimental): 200ng GSK2445053
  Interventions: Drug: 200ng GSK2445053
- Part 1 Cohort 4 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 5 GSK245053 (Experimental): 400ng GSK2445053
  Interventions: Drug: 400ng GSK2445053
- Part 1 Cohort 5 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 6 GSK2445053 (Experimental): 1000ng GSK2245053
  Interventions: Drug: 1000ng GSK2445053
- Part 1 Cohort 6 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 7 GSK2445053 (Experimental): 2000ng GSK2445053
  Interventions: Drug: 2000ng GSK2445053
- Part 1 Cohort 7 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Part 1 Cohort 8 GSK2445053 (Experimental): 4000ng GSK2445053
  Interventions: Drug: 4000ng GSK2445053
- Part 1 Cohort 8 Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2 ng GSK2445053 — 2ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 1 GSK2445053
Drug: 20ng GSK2445053 — 20ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 2 GSK2445053
Drug: 100ng GSK2445053 — 100ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 3 GSK2245053
Drug: 200ng GSK2445053 — 200ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 4 GSK2445053
Drug: 400ng GSK2445053 — 400ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 5 GSK245053
Drug: 1000ng GSK2445053 — 1000ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 6 GSK2445053
Drug: 2000ng GSK2445053 — 2000ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 7 GSK2445053
Drug: 4000ng GSK2445053 — 4000ng GSK2445053 administered intranasally
  Arms: Part 1 Cohort 8 GSK2445053
Drug: Placebo — Placebo administered intranasally
  Arms: Part 1 Cohort 1 Placebo; Part 1 Cohort 2 Placebo; Part 1 Cohort 3 Placebo; Part 1 Cohort 4 Placebo; Part 1 Cohort 5 Placebo; Part 1 Cohort 6 Placebo; Part 1 Cohort 7 Placebo; Part 1 Cohort 8 Placebo

SUMMARY:
GSK2245035 is a highly selective Toll-like Receptor 7(TLR7) agonist capable of preferentially inducing the production of interferon alpha (IFNα) versus tumor necrosis factor alpha (TNFα). The aim of this FTIH study is to collect tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) information to enable the identification of appropriate safe doses of intranasal (i.n) GSK2245035, associated with up-regulation of TLR7-mediated genes in the nasal milieu, for use in subsequent clinical drug development studies. There will be two parts to the study: Healthy Volunteers will be dosed in escalating single doses in Part 1, followed by Allergic Rhinitis (AR) subjects dosed similarly in Part 2.

DETAILED DESCRIPTION:
This is a First Time in Human (FTIH) study to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single, escalating doses of intranasal (i.n.) GSK2245035 in healthy male volunteers (HVT) and male subjects with allergic rhinitis (AR). The safety and tolerability of single i.n. GSK2245035 dosing will be assessed and established in HVT before the initiation of evaluation in AR.

GSK2245035 is a highly selective Toll-like Receptor 7 (TLR7) agonist capable of preferentially inducing the production of IFNα rather than TNFα. Activation of TLR7 is known to result in upregulation of co-stimulatory signals on antigen-presenting cells and in generation of pro-inflammatory mediators that can shift bystander immune responses towards a Helper T-cell Type 1/ Regulatory T cell (Th1/Treg) phenotype and therefore reduce the magnitude of Helper T-cell Type 2 (Th2) reactivity. In this context, it is proposed that i.n. GSK2245035 administration may alter the airways immune environment in a way that results in long-lasting control of AR symptoms and potentially disease remission through persistent modification of the underlying aberrant Th2 responsiveness to aeroallergens.

The aim of this study is to collect tolerability, PK and PD information to enable the identification of appropriate safe doses of i.n. GSK2245035, associated with up-regulation of TLR7-mediated genes in the nasal milieu, for use in subsequent clinical drug development studies. The study will be divided in to two parts. Part 1, involving only healthy volunteers, will consist of 8 cohorts receiving doses from 2 nanograms (2 ng) to 4000ng or a placebo dose. Administration within each cohort will be staggered so that two subjects (one receiving drug and one placebo) will be dosed and monitored for 24 hours before any subsequent doses.

Screening for part 2 of the study will begin once data from cohort 4 in part 1 has been found to be satisfactory. Part 2 will involve subjects with Allergic Rhinitis and be divided into three cohorts receiving doses between 20ng and 4000ng or a placebo dose.

ELIGIBILITY:
Inclusion Criteria for all subjects (parts 1 and 2)

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history,physical examination, laboratory testsand cardiac monitoring. A subject with a clinical abnormality or laboratoryparameters outside the reference range for the population being studied may be included only if the Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1 of the protocol. This criterion must be followed from the time of the first dose of study medication until one week post-dosing.
* Body weight greater than or equal to 50 kilograms (kg) and Body Mass Index (BMI) within the range 19 - 29.9 kilograms per square metre (kg/m2) inclusive.
* 12 lead Electrocardiogram without any clinically significant abnormality as judged by the Investigator, and average QT interval (QTc), QT interval corrected for Basett (QTcB) or QT interval corrected for Fredericia (QTcF) less than 450 milliseconds
* Aspartate transaminase (AST), alanine transamine (ALT), alkaline phosphatase and bilirubin less than 1.5 x Upper Limit of Normal (ULN) (isolated bilirubin greater than1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Subjects have a screening pre-challenge Forced Expiratory Volume in 1 second (FEV1) greater than or equal to 80% and a baseline FEV1/FVC greater than or equal to 70% of the predicted value.
* Subjects should refrain from smoking between screening and the end of the study, and have a negative test for cotinine/ carbon monoxide (CO) at pre-dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all the required study measurements.

Inclusion Criteria for Allergic Rhinitics only (Part 2)

* History and diagnosis of symptomatic seasonal allergic rhinitis to pollen, for more than 3 years.
* Positive skin allergy test (wheal greater than or equal to 4miliimetres) or radioallergosorbent test (RAST) greater than or equal to Class 2, for pollen allergens.
* Subjects have a Total Nasal Symptom Score (TNSS) score of greater than or equal to 3 during the current pollen season (Total nasal symptom score is the sum of nasal congestion, rhinorrhoea, nasal itch and sneeze, each of which are scored on a scale from 0 to 3).

Exclusion Criteria for all subjects (Parts 1 and 2):

* History of immunologic or haematologic deficiencies or diseases, except conditions that in the opinion of the Investigator and the GSK Medical Monitor are unlikely to introduce additional risk factors.
* Current diagnosis of asthma.
* Nasal conditions likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, other nasal malformations or history of frequent nosebleeds.
* History of haematologic, gastro-intestinal, hepatic, renal or other condition that may influence the absorption, distribution, metabolism, excretion or action of the drug.
* History of frequent headaches and/or migraine.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for Human Immunodeficiency Virus antibody
* A positive screening or pre-dose drug/alcohol screen, or a positive pre-dose smoking test
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 grams (8g) of alcohol: a half-pint or approximately 240 millilitres (240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within 3 months prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 6 months prior to the first dosing day.
* History of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates participation in this study.
* Donation of blood or blood products in excess of 500 mL within a 90-day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated

Exclusion Criteria for healthy volunteers only (part 1)

* History of rhinitis, including allergic, non-allergic rhinitis and rhinosinusitis. Subjects with recent upper respiratory tract infections (URTIs) will be allowed in the study only if their nasal symptoms have been completely resolved for more than 3 weeks prior to screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to entry to the clinic, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Exclusion criteria for Allergic Rhinitics only (part 2)

* Subjects with recent upper respiratory tract infections (URTIs) will be allowed in the study only if their nasal symptoms have been completely resolved for more than 3 weeks prior to screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to entry into the clinic, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Subjects using treatment for allergies and AR may participate in the study if they remain free of medication for the following periods of time prior to entry into the clinic:

  * Nasal antihistamines: 48 hours
  * Oral antihistamines A (cetirizine, fexofenadine, loratadine, desloratadine): 72 hours
  * Oral antihistamines B (all others): 72 hours
  * Nasal decongestants: 24 hours
  * Oral decongestants: 24 hours
  * Nasal glucocorticosteroids: 4 weeks
  * Oral glucocorticosteroids: 12 weeks
  * Oral leukotriene receptor antagonists: 7 days

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05-30 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
Safety | From screening until follow-up
  General safety endpoints, including AEs, vital signs, 12-lead ECG, body temperature and clinical laboratory safety tests to evaluate the safety and nasal tolerability of single escalation doses of GSK2245035 in healthy volunteers and individuals with Allergic Rhinitis.
Nasal Tolerability | From screening until follow-up
  Nasal examination and nasal symptom to assess nasal tolerability of single escalating doses of GSK2245035 in subjects with Allergic Rhinitis
TLR7-associated Biomarkers | From pre-dose until 3 days post-dose
  Evaluation of the induction of TLR7-induced blood biomarkers in the nasal lavage and nasal tissues of individuals with AR following single GSK2245035 administration versus placebo.

SECONDARY OUTCOMES:
Systemic PK | From pre-dose until 3 days post-dose
  Standard single dose derived plasma PK parameters for GSK2245035 in healthy volunteers and individuals with Allergic Rhinitis
Correlation Evaluation | From pre-dose until 3 days post-dose
  To evaluate the correlation between GSK2245035 dose - systemic PK - PD blood biomarkers - PD nasal biomarkers in healthy volunteer and subjects with Allergic Rhinitis.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tsitoura D, Ambery C, Price M, Powley W, Garthside S, Biggadike K, Quint D. Early clinical evaluation of the intranasal TLR7 agonist GSK2245035: Use of translational biomarkers to guide dosing and confirm target engagement. Clin Pharmacol Ther. 2015 Oct;98(4):369-80. doi: 10.1002/cpt.157. PMID 26044169
- See also: Results for study 114450 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114450?search=study&search_terms=114450#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114450 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register